CLINICAL TRIAL: NCT01854996
Title: A Phase I, Randomized, Single-Dose Study To Determine The Relative Bioavailability Of Capsule Vs Oral Dispersion And The Effect Of Food On The Pharmacokinetics Of Orally Administered PF-05089771 As Capsule In Healthy Volunteers
Brief Title: Relative Bioavailability With PF-05089771 Capsule Versus Oral Dispersion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B3291020
Record Dates: First submitted 2013-05-08; First posted 2013-05-16 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
MeSH Terms: interventions — PF-05089771

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oral disperion fasted (Experimental): A single dose of 450 mg PF-05089771 TS oral dispersion in fasted conditions.
  Interventions: Drug: PF-05089771
- Capsule fasted (Experimental): single dose of 450 mg PF-05089771 TS as 3 x 150 mg capsules in fasted conditions
  Interventions: Drug: PF-05089771
- Capsule fed (Experimental): single dose of 450 mg PF-05089771 TS as 3 x 150 mg capsules in fed conditions
  Interventions: Drug: PF-05089771

INTERVENTIONS:
Drug: PF-05089771 — 450mg
  Other Names: no specified
  Arms: Oral disperion fasted
Drug: PF-05089771 — 450mg
  Other Names: no specified
  Arms: Capsule fasted
Drug: PF-05089771 — 450mg
  Other Names: no specified
  Arms: Capsule fed

SUMMARY:
This study aims to test plasma exposure to PF-05089771 with same formulation will be used for phase II trials (capsule).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests). Females must be of non-childbearing potential.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* An informed consent document signed and dated by the subject or a legally acceptable representative, indicating that the subject has been informed of all pertinent aspects of the trial.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal (i.e recurrent uric nephrolithiasis), endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 48 hours
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 48 hours

SECONDARY OUTCOMES:
Number of Participants With Laboratory Test Values of Potential Clinical Importance | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291020&StudyName=Relative%20Bioavailability%20with%20PF-05089771%20Capsule%20Versus%20Oral%20Dispersion